CLINICAL TRIAL: NCT03399136
Title: Fitness and Longevity in Exercise
Acronym: FLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, KrisAnn Oursler, Physician, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HP-00042601
Record Dates: First submitted 2018-01-04; First posted 2018-01-16 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: HIV-1-infection; Aging
Keywords: Exercise training; Intervention; Aerobic capacity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity aerobic exercise (Experimental): In the moderate-intensity aerobic exercise group, participants performed a self-paced 1-mile walk (3-5 METs) on an indoor track in the same exercise center as the high-intensity exercise group. Initial sessions lasted 20-30 minutes and were increased weekly to 45 minutes in parallel to the duration of the high-intensity exercise group.
  Interventions: Behavioral: Exercise training
- High-intensity aerobic exercise (Experimental): In the high-intensity aerobic exercise group, exercise training was performed on a motorized treadmill with occasional substitution with the elliptical machine as needed for joint pain. Target heart rate was based on the baseline treadmill test and was calculated as percentage of the heart rate reserve (HRR=maximal HR-resting HR). Initially, participants trained for 20-30 minutes at 50-60% of HRR. Duration and intensity was increased by 10% weekly so that within 5-7 weeks the aerobic exercise sessions lasted 30-45 minutes at 70-85% of HRR and at the end of the 16 weeks lasted 40-45 minutes at 75-90% of HRR.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Participants attended center-based exercise sessions three times per week at the research exercise training facility located at the Baltimore VA Medical Center. All exercise training was performed under the supervision of research exercise physiologists. Heart rate (HR) was measured continuously during each session using a Polar HR watch and chest strap allowing for assessment and maintenance of treatment fidelity. Exercise logs included details on exercise type, duration, time in target heart rate zone, blood pressure and perceived intensity during each training session.

SUMMARY:
The study objective was to determine the safety and efficacy of aerobic exercise in older HIV-infected men in a randomized trial comparing different levels of exercise intensity.

DETAILED DESCRIPTION:
The study was a randomized trial of moderate-intensity versus high-intensity aerobic exercise (AEX) training in older HIV-infected adults. Funding was provided by K23 AG024896 (PI, Oursler) and the UMB Claude D. Pepper Older Americans Independence Center P60 AG12583 (PI, Goldberg).

The central hypothesis was that high-intensity AEX training is well-tolerated and significantly increases aerobic capacity in older HIV-infected adults.

The study met its objectives:

1. Scientific AIMS met:

   1. High-intensity AEX training significantly increases aerobic capacity
   2. Both moderate-intensity and high-intensity AEX training improve ambulatory function and endurance.
   3. Activity of skeletal muscle oxidative enzymes is reduced, and associated with aerobic capacity.
2. Feasibility Objectives met:

   1. AEX training is safe and well-tolerated in older HIV-infected adults.
   2. Skeletal muscle punch biopsy is safe and well-tolerated in older HIV-infected adults.
   3. Preliminary data was collected on plasma biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* stable combination antiretroviral therapy (cART)

Exclusion Criteria:

* AIDS defining conditions in the prior six months
* Conditions that increase the risk of exercise training per the American College of Sports Medicine (ACSM)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-07-19 (Actual); Primary Completion 2010-10-29 (Actual); Study Completion 2012-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline Cardiorespiratory Fitness at 16 weeks | 16-weeks
  Cardiorespiratory Fitness measured by VO2peak

SECONDARY OUTCOMES:
Change from baseline Six-minute walk distance at 16 weeks | 16-weeks
  Distance walked at normal pace in 6 minutes
Change from baseline body composition at 16 weeks | 16-weeks
  body composition measured as total and regional lean tissue and fat mass (DXA)
Change from baseline exercise endurance at 16 weeks | 16-weeks
  exercise endurance measured as time on treadmill during modified Bruce protocol

OTHER OUTCOMES:
skeletal muscle oxidative function | baseline
  activity of enzymes in oxidative function from muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Krisann Oursler, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No
Data, which include PHI, are available from the University of Maryland School of Medicine Institutional Review Board for researchers who meet the criteria for access to confidential data.

REFERENCES:
- [Result] Ortmeyer HK, Ryan AS, Hafer-Macko C, Oursler KK. Skeletal muscle cellular metabolism in older HIV-infected men. Physiol Rep. 2016 May;4(9):e12794. doi: 10.14814/phy2.12794. PMID 27166139